CLINICAL TRIAL: NCT01887236
Title: The Effect of Exercise Training Programs: Step and Stability Ball on Balance and Obstacle Avoidance in Older People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HYMC-38-13
Record Dates: First submitted 2013-06-23; First posted 2013-06-26 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Aging

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Step Physical Activity (Active Comparator): A physical activity program that is based on the Step Apparatus Training Program
  Interventions: Behavioral: Step physical activity program
- Stability Ball (Active Comparator): A physical activity program that is based on the Stability Ball
  Interventions: Behavioral: Stability Ball Program

INTERVENTIONS:
Behavioral: Step physical activity program — Participants will take part in a biweekly, 8 week physical activity program that will include step exercises
  Arms: Step Physical Activity
Behavioral: Stability Ball Program — Participants will take part in a biweekly, 8 week physical activity program that will include stability ball exercises
  Arms: Stability Ball

SUMMARY:
Individuals of advanced age undergo both physical and cognitive deterioration. The aim of this study is to explore the effect of two types of physical activity on stability parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age above 65
* Able to undergo physical activity for 45 minutes twice a week

Exclusion Criteria:

* All Others

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Stability | 3 months
  Stability will be measured with the following tests:
  Timed Get Up and Go , One Leg Stand Test, Functional Reach Test,Tinetti Balance both before and after the 8 week physical activity program and the difference will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Zinman College for Physical Education and Sport Sciences, Netanya, Israel